CLINICAL TRIAL: NCT01570244
Title: An Open-label, Two-period, Fixed-sequence, Phase I Trial to Evaluate the Effect of Multiple Doses of 240 mg BI 201335 QD on the Multiple-dose Pharmacokinetics of a Combination of Ethinylestradiol and Levonorgestrel in Healthy Premenopausal Female Volunteers
Brief Title: Drug-drug Interaction of BI 201335 and Microgynon
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1220.56; 2011-006061-17 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Levonorgestrel; Ethinyl Estradiol; faldaprevir

ARMS (2):
- Reference (Experimental): multiple doses of Microgynon
  Interventions: Drug: levonorgestrel; Drug: Ethinylestradiol
- Test (Active Comparator): multiple doses of Microgynon + BI 201335
  Interventions: Drug: levonorgestrel; Drug: Ethinylestradiol; Drug: BI 201335

INTERVENTIONS:
Drug: levonorgestrel — multiple doses
  Arms: Test
Drug: Ethinylestradiol — multiple doses
  Arms: Test
Drug: levonorgestrel — multiple doses
  Arms: Reference
Drug: BI 201335 — multiple doses
  Arms: Test
Drug: Ethinylestradiol — multiple doses
  Arms: Reference

SUMMARY:
This study will investigate possible effect of multiple oral doses of BI 201335 on the steady state pharmacokinetics of ethinylestradiol and levonogestrel

ELIGIBILITY:
Inclusion criteria:

1. Healthy female subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1220.56.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

REFERENCES:
- [Derived] Sabo JP, Lang B, Elgadi M, Huang F. Effect of the hepatitis C virus protease inhibitor faldaprevir on the pharmacokinetics of an oral contraceptive containing ethinylestradiol and levonorgestrel in healthy female volunteers. Antimicrob Agents Chemother. 2015 Jan;59(1):514-9. doi: 10.1128/AAC.03589-14. Epub 2014 Nov 10. PMID 25385099

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: The trial was a nonrandomised, noncontrolled, open-label, 2-period fixed-sequence trial to evaluate the possible effect of multiple doses of faldaprevir on the multiple-dose pharmacokinetics of a combination of ethinylestradiol and levonorgestrel. The trial was to be performed in 16 healthy female volunteers.
  Period 1: Microgynon (150 μg Ethinylestradiol+30 μg Levonorgestrel) tablets.
  Period 2: Microgynon tablets and Faldaprevir.
Period: Microgynon
Arm/Group | All Subjects
Started | 16
Completed | 16
Not Completed | 0
Period: Microgynon+Faldaprevir
Arm/Group | All Subjects
Started | 16
Completed | 15
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: The trial was a nonrandomised, noncontrolled, open-label, 2-period fixed-sequence trial to evaluate the possible effect of multiple doses of faldaprevir on the multiple-dose pharmacokinetics of a combination of ethinylestradiol and levonorgestrel. The trial was to be performed in 16 healthy female volunteers.
Arm/Group | All Subjects
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: AUCt,ss of Ethinylestradiol
Description: Area under the curve over the dosing interval t under steady state conditions of ethinylestradiol
Time Frame: on day 13 of first period and on day 8 of second period 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 hours (h) after drug administration
Population: Pharmacokinetic (PK) set: all subjects in the treated set who provided at least 1 observation for at least 1 primary pharmacokinetic endpoint, who did not have important protocol violations relevant to the evaluation of PK endpoints, and who did not have vomiting until 2·median tmax,ss of ethinylestradiol or levonorgestrel on Day 13 or on Day 8.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Groups:
- Microgynon: Multiple doses of Microgynon (150 µg Ethinylestradiol+30 µg Levonorgestrel) tablets once daily in the morning.
- Microgynon + Faldaprevir: Multiple doses of Microgynon (150 µg Ethinylestradiol+30 µg Levonorgestrel) tablets once daily in the morning.
  Faldaprevir: loading dose of 480 mg (morning and evening doses of 240 mg on Day 1 of Period 2), on subsequent days 240 mg once daily in the morning.
Arm/Group | Microgynon | Microgynon + Faldaprevir
Number analyzed (Participants) | 16 | 15
pg*h/mL | 1010 (23.5) | 1450 (27.8)
Statistical Analysis 1: Comparison: Microgynon vs Microgynon + Faldaprevir; relative bioavailability comparison (Microgynon + Faldaprevir : Microgynon) of Ethinylestradiol; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 140.96, 90% CI 2-sided [133.84 to 148.47], Standard Deviation 8.1 — the standard deviation is actually the geometric coefficient of variation

2. Primary Outcome: Cmax,ss of Ethinylestradiol
Description: maximum measured concentration over the uniform dosing interval under steady state conditions of ethinylestradiol
Time Frame: on day 13 of first period and on day 8 of second period 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 h after drug administration
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Microgynon | Microgynon + Faldaprevir
Number analyzed (Participants) | 16 | 15
pg/mL | 108 (23.6) | 127 (25.1)
Statistical Analysis 1: Comparison: Microgynon vs Microgynon + Faldaprevir; relative bioavailability comparison (Microgynon + Faldaprevir : Microgynon) of Ethinylestradiol; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Odds Ratio (OR) = 114.82, 90% CI 2-sided [105.49 to 124.97], Standard Deviation 13.2 — the standard deviation is actually the geometric coefficient of variation

3. Primary Outcome: C24,ss of Ethinylestradiol
Description: measured concentration of the analyte at the end of dosing interval under steady state conditions of ethinylestradiol
Time Frame: as for outcome 2
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Microgynon | Microgynon + Faldaprevir
Number analyzed (Participants) | 16 | 15
pg/mL | 19.1 (32.9) | 33.2 (42.9)
Statistical Analysis 1: Comparison: Microgynon vs Microgynon + Faldaprevir; relative bioavailability comparison (Microgynon + Faldaprevir : Microgynon) of Ethinylestradiol; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 171.37, 90% CI 2-sided [160.20 to 183.33], Standard Deviation 10.5 — the standard deviation is actually the geometric coefficient of variation

4. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Physical Examination, Blood Chemistry, Haematology, Urinanalysis and ECG.
Description: Clinical relevant abnormalities for Vital Signs, Physical Examination, Blood Chemistry, Haematology, Urinanalysis and ECG. New abnormal findings or worsening of baseline conditions were reported as Adverse Events.
Time Frame: from drug administration up to 14 days
Population: Treated set: This subject set included all 16 subjects who were administered trial medication and were documented to have taken at least 1 dose of investigational treatment.
Measure: Number; unit: participants
Arm/Group | Microgynon | Microgynon + Faldaprevir
Number analyzed (Participants) | 16 | 16
participants | 0 | 0

5. Secondary Outcome: Number of Participants With Drug Related Adverse Events
Description: number of participants with investigator-defined drug related adverse events
Time Frame: from drug administration up to 14 days
Population: treated set
Measure: Number; unit: participants
Arm/Group | Microgynon | Microgynon + Faldaprevir
Number analyzed (Participants) | 16 | 16
participants | 2 | 15

6. Primary Outcome: AUCτ,ss of Levonorgestrel
Description: Area under the curve over the dosing interval τ under steady state conditions of levonorgestrel
Time Frame: as for outcome 2
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Microgynon | Microgynon + Faldaprevir
Number analyzed (Participants) | 16 | 15
ng*h/mL | 83.3 (42.0) | 120 (40.6)
Statistical Analysis 1: Comparison: Microgynon vs Microgynon + Faldaprevir; relative bioavailability comparison (Microgynon + Faldaprevir : Microgynon) of Levonorgestrel; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric mean ratio = 140.53, 90% CI 2-sided [136.40 to 144.78], Standard Deviation 4.6 — the standard deviation is actually the geometric coefficient of variation

7. Primary Outcome: Cmax,ss of Levonorgestrel
Description: maximum measured concentration over the uniform dosing interval under steady state conditions of levonorgestrel
Time Frame: as for outcome 2
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Microgynon | Microgynon + Faldaprevir
Number analyzed (Participants) | 16 | 15
ng/mL | 7.57 (34.9) | 8.95 (33.3)
Statistical Analysis 1: Comparison: Microgynon vs Microgynon + Faldaprevir; relative bioavailability comparison (Microgynon + Faldaprevir : Microgynon) of Levonorgestrel; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 115.28, 90% CI 2-sided [110.81 to 119.92], Standard Deviation 6.1 — the standard deviation is actually the geometric coefficient of variation

8. Primary Outcome: C24,ss of Levonorgestrel
Description: measured concentration of the analyte at the end of dosing interval under steady state conditions of levonorgestrel
Time Frame: as for outcome 2
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Microgynon | Microgynon + Faldaprevir
Number analyzed (Participants) | 16 | 15
ng/mL | 2.43 (49.4) | 3.85 (47.9)
Statistical Analysis 1: Comparison: Microgynon vs Microgynon + Faldaprevir; relative bioavailability comparison (Microgynon + Faldaprevir : Microgynon) of Levonorgestrel; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 153.85, 90% CI 2-sided [145.99 to 162.14], Standard Deviation 8.2 — the standard deviation is actually the geometric coefficient of variation

ADVERSE EVENTS:
Time Frame: from the time the subject signed the informed consent (56 to 28 days before drug administration) through the observational phase until the end-of-study examination (6 to 14 days after the end of period 2)
Description: During the run-in-period, the volunteers were to be contacted at least twice and asked to report adverse events and concomitant medication. In addition, each volunteer was to be assessed regularly by the medical staff throughout the clinical trial as well as at the end of observation and whenever necessary as deemed by the investigator.
Groups:
- Microgynon + BI 201335: Multiple doses of Microgynon (150 µg Ethinylestradiol+30 µg Levonorgestrel) tablets once daily in the morning.
  Faldaprevir: loading dose of 480 mg (morning and evening doses of 240 mg on Day 1 of Period 2), on subsequent days 240 mg once daily in the morning.
Arm/Group | Microgynon | Microgynon + BI 201335
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 12/16 | 14/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Microgynon (N=16) | Microgynon + BI 201335 (N=16)
Tachycardia (Cardiac disorders) | 0 | 1
Ocular icterus (Eye disorders) | 0 | 6
Abdominal discomfort (Gastrointestinal disorders) | 0 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 8
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 4
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Swelling (General disorders) | 1 | 0
Oral herpes (Infections and infestations) | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 7
Increased appetite (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 3
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 5 | 6
Orthostatic intolerance (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Apathy (Psychiatric disorders) | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.